CLINICAL TRIAL: NCT06404957
Title: The Effect of Mindfulness-based Nursing Interventions Applied to Hemodialysis Patients on Psychosocial Adaptation
Brief Title: Effect of Mindfulness-based Applied to Hemodialysis Patients on Psychosocial Adaptation
Acronym: EMBAHPPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, GÜLGÜNDURAT, Associate professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SakaryaU-Hemodialysis
Record Dates: First submitted 2022-12-22; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis; Psychosocial Adaptation
Keywords: Mindfulness; Hemodialysis; Nursing; Psychosocial Adaptation

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Applied (Experimental): Patients in the experimental group were determined, 6-week, 90-minute-a-week mindfulness-based nursing interventions were taught, and group applications were made before the intervention and after; pre-test and post-test questionnaires were applied.
  Interventions: Behavioral: Mindfulness-based Applied
- Control groups (Active Comparator): No intervention was made in the control group. At the start of the intervention step of the study and after six weeks, pre-test and post-test questionnaires were applied to control groups.
  Interventions: Behavioral: Active Comparator: Control groups

INTERVENTIONS:
Behavioral: Mindfulness-based Applied — Mindfulness-Based Practices is planned to be an 8-week program of mindfulness meditation and gentle Hatha yoga taught in an online class for up to 14 participants.
  Arms: Mindfulness-based Applied
Behavioral: Active Comparator: Control groups — No intervention will be made in this group.
  Arms: Control groups

SUMMARY:
The goal of this clinical study is to adapt mindfulness-based nursing interventions to hemodialysis patients and to investigate their effects on their psychosocial adjustment.

The main question[s] it aims to answer are:

Do consciously applied nursing interventions increase the psychosocial adjustment to the disease in hemodialysis patients? Do mindfulness-based nursing interventions increase body and mind awareness in hemodialysis patients? Researchers will compare the experimental and control groups to see if mindfulness-based interventions have an effect on the psycho-social adjustment of hemodialysis patients.

DETAILED DESCRIPTION:
Primary Aims Test the efficacy of an adapted Mindfulness-Based Stress Reduction program to reduce symptoms and improve psychosocial adaption by 6 weeks.

Hypotheses

Primary: The mindfulness-based program increases the psychosocial adjustment to the disease in hemodialysis patients.

Secondary: Mindfulness-based program increases body and mind awareness in hemodialysis patients.

Long-range Goal: To develop evidence-based recommendations for non-pharmacologic strategies that provide psychosocial adaptation relief to hemodialysis patients and are safe, practical, and cost-effective.

Interventions: The Mindfulness-based Applied program includes the curricular content of the standard 6 week. A trained teacher provides instruction in meditation techniques, including body scan, standing, sitting, and walking meditations, and mindful yoga.

The attention control consists of 90-minute online workshops. Audio recordings and written materials related to awareness exercises will be given to the participants at the end of each session so that they can do home practices.

Recruiting Methods:

It will consist of hemodialysis patients receiving service from hemodialysis centers located in a province in the west of Turkey. The sample of the study will consist of individuals who voluntarily agree to participate in the study and who comply with the research criteria.

Data Collection Tools Mindfulness scale: Mindful Awareness Attention Scale (MAAS) The psychosocial adjustment to illness scale (PAIS-SR) Hemodialysis Stressor Scale (HSS)

Study Design: Randomized controlled experimental study

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis treatment
* Between the ages of 18-65

Exclusion Criteria:

* Patients with acute renal failure
* Current hospitalization, current ongoing chemotherapy or radiotherapy
* Cognitive dysfunction or mental retardation
* Current substance abuse
* Entering hemodialysis due to current psychotropic drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Mindfulness-Based Practice Applied to Hemodialysis Patients | 6 weeks
  Awareness-Based Practice Applied to Haemodialysis Patients is expected to affect the psychosocial adaptation of patients to their diseases.. Psychosocial Adjustment to Illness Self-Report Scale (PAIS-SR) was used to assess this outcome measure. Each item is scored on a scale ranging from 0 to 3. Largely negative differences since the disease are evaluated with a score of 3 and positive differences with a score of 0. In studies conducted with PAIS-SR, scores lower than 35 are evaluated as good psychosocial adjustment, scores between 35-51 as moderately good psychosocial adjustment, and scores higher than 51 as poor adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Şen Tepe, MSc, Principal Investigator — Sakarya University Faculty of Healt Science; Gülgün Durat, Assoc. Prof., Study Director — Sakarya University Faculty of Healt Science
Locations (1):
- Çiğdem Şen Tepe, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sohn BK, Oh YK, Choi JS, Song J, Lim A, Lee JP, An JN, Choi HJ, Hwang JY, Jung HY, Lee JY, Lim CS. Effectiveness of group cognitive behavioral therapy with mindfulness in end-stage renal disease hemodialysis patients. Kidney Res Clin Pract. 2018 Mar;37(1):77-84. doi: 10.23876/j.krcp.2018.37.1.77. Epub 2018 Mar 31. PMID 29629280
- [Background] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293
- [Background] Gross CR, Reilly-Spong M, Park T, Zhao R, Gurvich OV, Ibrahim HN. Telephone-adapted Mindfulness-based Stress Reduction (tMBSR) for patients awaiting kidney transplantation. Contemp Clin Trials. 2017 Jun;57:37-43. doi: 10.1016/j.cct.2017.03.014. Epub 2017 Mar 22. PMID 28342990
- See also: Turkish Society of Nephrology Registry 2019 — https://nefroloji.org.tr/uploads/folders/file/registry_2019.pdf